CLINICAL TRIAL: NCT05620329
Title: University of North Carolina Pleural Fluid Registry
Brief Title: UNC Pleural Fluid Registry
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1754
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; Lung Infection; Breast Cancer; Malignant Pleural Effusion; Empyema
Keywords: biospecimen; pleural fluid; lung cancer; cancer; infection; breast cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Pleural Effusion, Malignant; Empyema; Neoplasms; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 32 Years
Biospecimen Retention: Samples With DNA — Blood and pleural fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pleural Fluid Registry: Any subject who has pleural fluid buildup from lung cancer, breast cancer, or lung infection

SUMMARY:
Research with biospecimens such as blood, tissue, or body fluids can help researchers understand how the human body works. Researchers can make new tests to find diseases, understand how treatments work, or find new ways to treat a disease. The purpose of this study is to collect biospecimens for research from patients with known or suspected lung cancer. The information learned from the biospecimens may be used in future treatments. The purpose of this protocol is to create a pleural fluid registry for use in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older
* Inpatients and outpatients
* Diagnosed with pleural fluid, are referred for and undergo clinically indicated drainage who have clinical evidence of:
* pulmonary infection (such as fever, leukocytosis, new or worsening infiltrate on chest x-ray, or clinical deterioration) with effusion
* malignancy

Exclusion Criteria:

* A subject will not be eligible for inclusion in this registry if, in the investigator's (or treating clinician's) opinion, the patient has any concurrent medical condition that may preclude their ability to undergo pleural fluid drainage safely.
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC patients
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2050-01-24 (Estimated); Study Completion 2050-01-24 (Estimated)

PRIMARY OUTCOMES:
Creation of a pleural fluid registry | 32 years
  Biological specimens and corresponding clinical data from subjects will be collected during standard of care procedures and medical record abstraction to support the creation of a pleural fluid registry.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Akulian, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lingeberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials